CLINICAL TRIAL: NCT07334600
Title: The Effect of 1% Andaliman Fruit Extract Cream (Zanthoxylum Acanthopodium DC.) on Seborrheic Keratosis
Brief Title: Effect of 1% Andaliman Fruit Extract Cream on Facial Seborrheic Keratosis
Acronym: ANDAL-SK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitas Sumatera Utara (Other)
Responsible Party: Principal Investigator, Sri Nauli Dewi Lubis, Departement of Dermatology and Venereology, Faculty of Medicine, Universitas Sumatera Utara, Medan, Indonesia, Universitas Sumatera Utara
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: USU-DV-SK-AND-2025; No.66/KEPK/USU/2025 (Other: Health Research Ethics Committee, Faculty of Medicine, Universitas Sumatera Utara)
Record Dates: First submitted 2025-12-30; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Seborrheic Keratosis
Keywords: Andaliman; Zanthoxylum acanthopodium; Topical herbal therapy; Facial skin lesions; Benign skin tumor
MeSH Terms: conditions — Keratosis, Seborrheic

STUDY DESIGN:
Intervention Model Description: This study used a single-arm, one-group pretest-posttest design in which all participants received the same topical intervention and were evaluated before and after treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Andaliman 1% Cream (Experimental): Participants in this single-arm study received topical treatment with 1% andaliman fruit extract cream (Zanthoxylum acanthopodium DC.). The cream was applied to facial seborrheic keratosis lesions for a treatment period of 12 weeks, with clinical evaluations performed at baseline and during follow-up visits.
  Interventions: Other: 1% Andaliman Fruit Extract Cream

INTERVENTIONS:
Other: 1% Andaliman Fruit Extract Cream — This intervention consisted of a topical cream containing 1% andaliman (Zanthoxylum acanthopodium DC.) fruit extract. Participants applied the cream directly to facial seborrheic keratosis lesions for a period of 12 weeks. The treatment was administered as a single intervention without a comparator, and participants were monitored for clinical response, safety, and adherence throughout the study period.
  Other Names: Zanthoxylum acanthopodium DC. Extract Cream

SUMMARY:
Seborrheic keratosis is a common benign skin growth that often appears on the face and may cause cosmetic concerns. This study aimed to evaluate the effectiveness and safety of a 1% andaliman fruit extract cream (Zanthoxylum acanthopodium DC.) as a topical treatment for facial seborrheic keratosis.

The study used a one-group pretest-posttest design and involved adult patients with seborrheic keratosis who received the cream for 12 weeks. Changes in lesion size were measured over time, and participants were monitored for side effects and overall satisfaction. The results of this study are expected to provide evidence on the potential use of a natural topical therapy for improving the appearance of seborrheic keratosis.

DETAILED DESCRIPTION:
This study was a quasi-experimental clinical trial using a one-group pretest-posttest design to evaluate the effect of a 1% andaliman fruit extract cream (Zanthoxylum acanthopodium DC.) on seborrheic keratosis lesions. The study was conducted at the Outpatient Clinic of UPT Puskesmas Padang Bulan, Medan, Indonesia.

Ethical approval was obtained from the Health Research Ethics Committee of Universitas Sumatera Utara (Approval No. 66/KEPK/USU/2025), and authorization was granted by the Research Division of the North Sumatra Provincial Health Office. Written informed consent was obtained from all participants prior to enrollment.

Eligible participants were adults aged 18 to 50 years with clinically and dermoscopically diagnosed common seborrheic keratosis lesions located on the facial region. Participants applied a 1% andaliman fruit extract cream to the lesion area and were followed for 12 weeks. Lesion size was measured at baseline and during follow-up visits to assess treatment response.

Participants were excluded if they were pregnant or breastfeeding, had used topical treatments such as 5-fluorouracil, retinoids, chemical peeling, laser therapy, or systemic or topical antioxidants prior to enrollment. Participants were considered dropouts if they did not comply with treatment instructions, used additional therapies during the study period, or discontinued treatment before completion.

The primary outcome of the study was the change in lesion size over time, while secondary observations included safety and patient satisfaction with the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-50 years.
* Patients diagnosed with common seborrheic keratosis lesions located on the facial region.
* Diagnosis confirmed by clinical and dermoscopic examination.
* Willing to participate in the study and provide written informed consent.

Exclusion Criteria:

* Pregnant or breastfeeding women.
* Use of topical treatments such as 5-fluorouracil, tretinoin, adapalene, glycolic acid, alpha-hydroxy acid, or antioxidants prior to enrollment.
* History of chemical peeling or laser therapy before enrollment.
* Use of oral or injectable antioxidants before or during the study period.
* Non-compliance with study procedures or use of additional therapies during the study period.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
Dermoscopic Changes of Seborrheic Keratosis Lesions | Baseline and Week 12
  Changes in dermoscopic features of seborrheic keratosis lesions before and after treatment with 1% andaliman fruit extract cream.

CONTACTS AND LOCATIONS:
Overall Officials: Imam Budi Putra, MD, Principal Investigator — Prof. Dr. Chairuddin Panusunan Lubis Universitas Sumatera Utara Hospital, Medan, Indonesia
Locations (1):
- Outpatient Clinic, Prof. Dr. Chairuddin Panusunan Lubis Universitas Sumatera Utara Hospital, Medan, North Sumatra, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Adrian, Syahputra RA, Juwita NA, Astyka R, Lubis MF. Andaliman (Zanthoxylum acanthopodium DC.) a herbal medicine from North Sumatera, Indonesia: Phytochemical and pharmacological review. Heliyon. 2023 May 12;9(5):e16159. doi: 10.1016/j.heliyon.2023.e16159. eCollection 2023 May. PMID 37251868
- [Background] Sepriani O, Nirhamidah N, Handayani D. Potensi ekstrak andaliman (Zanthoxylum acanthopodium DC.) sebagai antibakteri. ALOTROP. 2020.
- [Background] Chen L, Hu JY, Wang SQ. The role of antioxidants in photoprotection: a critical review. J Am Acad Dermatol. 2012 Nov;67(5):1013-24. doi: 10.1016/j.jaad.2012.02.009. Epub 2012 Mar 9. PMID 22406231
- [Background] James WD, Berger TG, Elston DM. Seborrheic keratosis. In: Andrews' Diseases of the Skin: Clinical Dermatology. 12th ed. Elsevier; 2016.
- [Background] Hafner C, Hartmann A, van Oers JM, Stoehr R, Zwarthoff EC, Hofstaedter F, Landthaler M, Vogt T. FGFR3 mutations in seborrheic keratoses are already present in flat lesions and associated with age and localization. Mod Pathol. 2007 Aug;20(8):895-903. doi: 10.1038/modpathol.3800837. Epub 2007 Jun 22. PMID 17585316
- [Background] Rajan A, Shukla P, Pai V. Role of dermoscopy in diagnosing and differentiating seborrheic keratoses. Egyptian Journal of Dermatology and Venereology. 2022.
- [Background] Klaassen KM. Treatment options for seborrheic keratosis. Dermatology Online Journal. 2018.
- [Background] Schwartz RA. Seborrheic keratosis: Clinical features and management. Journal of Dermatological Treatment. 2020.
- See also: General information about clinical trial registration and study protocol. — https://clinicaltrials.gov